CLINICAL TRIAL: NCT04064554
Title: A Prospective, Randomized, Open-label, Single-centered Clinical Study to Evaluate Safety and Immunogenicity of Bacillus Calmette-Guerin (BCG) Delivery Via Novel Micronjet600 Device Compared to Those Via Conventional Needle
Brief Title: Clinical Study to Evaluate Safety and Immunogenicity of Bacillus Calmette-Guerin (BCG) Delivery Via Novel Micronjet600 Device Compared to Those Via Conventional Needle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1-2017-0073
Record Dates: First submitted 2019-08-05; First posted 2019-08-22 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Tuberculosis; BCG Vaccination
Keywords: Tuberculosis; BCG vaccination
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: 1. Experimental: BCG vaccination with MicronJet600
  2. Comparator: BCG vaccination with conventional needle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MicronJet600 (Experimental): BCG vaccination with MicronJet600
  Interventions: Device: BCG vaccination with MicronJet600
- Conventional needle (Active Comparator): BCG vaccination with conventional needle
  Interventions: Device: BCG vaccination with conventional needle

INTERVENTIONS:
Device: BCG vaccination with MicronJet600 — BCG vaccination with MicronJet600
  Arms: MicronJet600
Device: BCG vaccination with conventional needle — BCG vaccination with conventional needle
  Arms: Conventional needle

SUMMARY:
The purpose of this study is to evaluate safety and immunogenicity of Bacillus Calmette-Guerin (BCG) delivery via Novel Micronjet600 device compared to those via conventional needle.

DETAILED DESCRIPTION:
This study is designed as prospective, randomized, open-label, single-centered. In this study, healthy adults who meet inclusion criteria will be randomized and receive a BCG vaccine either using a conventional needle or MicronJet600 device. After vaccination, adverse events and progress will be observed.

ELIGIBILITY:
Inclusion Criteria:

* 1) Subjects who voluntarily consented, after listening enough explanation for this study and the characteristics of medical devices and BCG vaccines.
* 2) Adults from 19 to 35 years
* 3) Tuberculin Skin Test negative
* 4) QFT-GIT(QuantiFERON-TB Gold In-Tube) Test negative
* 5) BMI from 19 to 35
* 6) A person who is determined to be suitable for the clinical trial as a result of the screening test.

(Even if the physical, laboratory, imaging, or electrocardiogram results are out of the normal range, the subject may participate if he or she has provided a clear basis for participation at the discretion of the investigator.)

Exclusion Criteria:

* 1) A person with a history of tuberculosis based on the medical history and chest radiograph, or who is suspected or confirmed to have a tuberculosis infection.
* 2) A person who has active fever except for mild acute upper respiratory infection or localized skin infection other than the site to be treated, or who has a fever of 38 °C or more within 1 week before application of the medical devices for the clinical trial.
* 3) A person who has not passed more than four weeks after the cure of virus infection (measles, mumps, chickenpox, and influenza).
* 4) A case that the subject has skin abrasions, open wounds, wounds, or scars on the site where the medical devices for the clinical trial.
* 5) A person who is unable to evaluate the local adverse effect because of tattoo, etc. on the site where the medical device for clinical trial is to be applied.
* 6) Patients with clinically significant arrhythmia difficult to participate in the clinical trial.
* 7) Patients with severe cardiac insufficiency (NYHA III and IV), a history of CABG(Coronary Artery Bypass Graft), and patients with cardiovascular diseases who are considered to be difficult to participate in the clinical trial.
* 8) A person with a known history of diabetes or a person whose diabetes was confirmed by a test.
* 9) Patients with hepatitis C or hepatitis B (in the case of hepatitis virus, healthy carriers may be participated at the discretion of the investigator) or positive for the serum test for human immunodeficiency virus (HIV).
* 10) Patients with severe immunosuppressive disease: congenital immunodeficiency such as severe combined immunodeficiency (SCID); leukemia; lymphoma, etc.
* 11) Patients with chronic renal insufficiency
* 12) A history of malignant tumors within 3 years excluding thyroid cancer (papillary, follicular, medullary types corresponding to Stage I or II), basal cell or squamous cell carcinoma on the skin, CIN(cervical intraepithelial neoplasia) and CIS(Carcinoma in situ) of the cervix, and intraepithelial carcinoma in other sites.
* 13) A case that a person has hypersensitivity or anamnesis for constitutivity constituting BCG.
* 14) Subjects who have not passed the predetermined period after receiving medication or treatment before the subjects participate in the clinical trial. (Refer to section 5.2.3.2)
* 15) Patients receiving concomitant medications (Refer to section 5.2.3.3)
* 16) A person who is unable to participate in the clinical trial period (about 6 months).
* 17) Patients scheduled for major surgery during the clinical trial.
* 18) A person who has a history of alcohol and other substance abuse for 6 months before screening.
* 19) Pregnant women or lactating women who are not willing to stop breastfeeding.
* 20) If the following are not applicable, (That is, you can only participate if):

  1. Women(female?) in the menopause (non-therapy-induced amenorrhea for more than 12 months)
  2. Infertility due to surgery (without ovaries and/or uterus)
  3. If the female subject have sexual intercourse with only one male partner who has been confirmed to have no semen after fertilization
  4. Female subjects who have agreed to abstinence during the clinical trial period

     * If the subject is assured of abstinence throughout the clinical trial period (only if abstinence is voluntarily selected by the subject and abstinence is consistent with the general lifestyle of the subject: e.g., Priest)

       * However, intermittent abstinence (e.g., ovulation, symptothermal method, or late ovulation) or external ejaculation is not a case of consent for abstinence.
  5. In the case of a woman who is in childbearing years, a woman who decides to use an effective method of contraception during the clinical trial period:

     * Oral contraception

       * Patch for contraception

         * Intrauterine Contraceptive Device (IUD)

           * Implant for contraception

             * Injection for contraception (Time-released type)

               * Hormone device in the uterus

                 * Tubal ligation and infertility surgery
* 21) Patient who has not passed 30 days since the date of signing the agreement of the previous clinical trial or who is currently participating in other clinical trial
* 22) Other diseases other than those listed above that the investigator deems inappropriate

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Visit 3(day 1, after vaccination) ~ Visit 6 (from 2 or 3 day of the Visit 5(day 85±7))
  Frequency and characteristics of adverse events after applying medical devices for clinical trials (aspect, materiality, results, etc.)
Adverse Events | during study period (Visit 3~Visit 6, 96 days)
  Frequency and characteristics of adverse events after applying medical devices for clinical trials (aspect, materiality, results, etc.)

SECONDARY OUTCOMES:
Average of usability VAS for medical device user | Visit 3 (day 1)
  The descriptive statistics (number of subjects, mean, standard deviation, median, minimum and maximum values) for the VAS(Visual Analogue Scale) scores measured at the time of the clinical device
  * VAS(visual analogue scale) :0(no paine)~10(wort possible, unbearable, excruciating pain).
  If necessary, a significance assessment will be performed through an independent t-test or Wilcoxon rank-sum test, and generalized linear model.
Spot Forming Unit (SFU) per PBMC(Peripheral Blood Mononuclear Cells) | Visit 1(day -28~2)
  Ex vivo IFN(Interferon) γ ELISpot analysis to measure the number of T cells that secrete cytokines by mycobacterial antigen-specific immune response
Spot Forming Unit (SFU) per PBMC | Visit 5(day 85±7)
  Ex vivo IFN γ ELISpot analysis to measure the number of T cells that secrete cytokines by mycobacterial antigen-specific immune response
Delta log10 CFU | Visit 1(day -28~2)
  Delta log 10 CFU at each time point evaluated by Ex vivo Mycobacterial Growth Inhibition Assay (MGIA). Delta log10 CFU=log(CFU count of each sample tube/CFU count of the growth control tube/incubation indays)
Delta log10 CFU | Visit 5(day 85±7)
  Delta log 10 CFU at each time point evaluated by Ex vivo Mycobacterial Growth Inhibition Assay (MGIA). Delta log10 CFU=log(CFU count of each sample tube/CFU count of the growth control tube/incubation indays)
Mycobacterial antigen specific T-cell | Visit 1(day -28~2)
  For intracellular cytokine staining (ICS) assay testing, the investigators will evaluate IFN-γ and TNF(Tumor Necrosis Factor)-α as intracellular cytokines. To assess ICS, blood samples were drawn before PPD(Purified protein derivative) administration at Visit 1. ICS assay will be performed using FACS(fluorescence activated cell sorting)(Fluorescence Activated Cell Sorting). The fraction of cells that are positive for any of cytokines measured at each point will be evaluated by total T cells, T4 and T8 subtype cells.
Mycobacterial antigen specific T-cell | Visit 5(day 85±7)
  For intracellular cytokine staining (ICS) assay testing, the investigators will evaluate IFN-γ and TNF-α as intracellular cytokines. To assess ICS, blood samples were drawn before PPD administration at Visit 5. ICS assay will be performed using FACS(Fluorescence Activated Cell Sorting). The fraction of cells that are positive for any of cytokines measured at each point will be evaluated by total T cells, T4 and T8 subtype cells.
PPD test result (positive or negative) after application of medical device for clinical trial | Visit 6 (from 2 or 3 day of the Visit 5(day 85±7))
  The number of test subjects who showed positive reactions at the time of evaluation (V6) will be presented for each group.
Diameter of induration (mm) or presence or absence of blister | Visit 6 (from 2 or 3 day of the Visit 5(day 85±7))
  Descriptive statistics (number of subjects, mean, standard deviation, median, minimum, and maximum values) for the diameter of the mandible measured at the time of administration of the medical device for clinical use are presented for each application group.
The diameter of the wheal | Visit 3 (day 1, after vaccination)
  The diameter of the wheal at the injection site immediately after BCG vaccination If necessary, a significance assessment will be performed through an independent t-test or Wilcoxon rank-sum test, and generalized linear model.
Fraction of subjects eligible for each grade in the injection fluid leakage assessment at the injection site | Visit 3 (day 1, immediately after vaccination)
  The number of test subjects to the degree of leakage assessment observed following the application of the clinical trial medical device will be presented for each application group. If necessary, a significance assessment will be performed through a chi-square test or Fisher's exact test.
Progress of normal reaction after BCG injection | Visit 3(day 1, after vaccination) ~ Visit 6 (from 2 or 3 day of the Visit 5(day 85±7))
  The normal reaction of the injected site observed after application of the medical device for clinical use will be indicated for each application group.
Diameter of the scar after BCG injection | Visit 3(day 1, after vaccination) ~ Visit 6 (from 2 or 3 day of the Visit 5(day 85±7))

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Yonsei University College of Medicine Division of Pulmonology, Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No